CLINICAL TRIAL: NCT07128342
Title: Use of Continuous Glucose Monitoring in Veterans With Uncontrolled Diabetes Managed Without Insulin Therapy
Brief Title: CGM Use in Non-insulin Patients With DM2
Acronym: CGM-DWI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milwaukee VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Carlos Mendez, Director, Diabetes Program, Milwaukee VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1856488
Record Dates: First submitted 2025-08-12; First posted 2025-08-18 (Actual); Last update posted 2025-08-18 (Actual); Status verified 2025-08

CONDITIONS: Diabetes; Type 2 Diabetes (T2DM); Obesity Type 2 Diabetes Mellitus; Non Insulin Dependent Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CGM group (Active Comparator): This group will receive CGM device for glucose monitoring
  Interventions: Device: CGM Group
- FSBG group (Active Comparator): This group will receive fingerstick device for glucose monitoring
  Interventions: Device: FSBG group

INTERVENTIONS:
Device: CGM Group — This group of patients will receive a CGM device to monitor their blood glucoses
  Arms: CGM group
Device: FSBG group — This group of patients will receive a fingerstick blood glucose (FSBG) device for glucose monitoring
  Arms: FSBG group

SUMMARY:
The U.S. Food and Drug Administration (FDA) has approved multiple Continuous Glucose Monitoring (CGM) devices from different manufacturers to be used as an aide in patients with type 1 and type 2 diabetes who require medications, and more recently, as over the counter versions for patients with and or without diabetes who want to better understand how diet and exercise may impact blood sugar levels. However robust evidence supporting that CGM is significantly superior to traditional home fingerstick blood glucose monitoring (FSBGM) in this population is lacking. Thus, Medicare and VHA only authorize use of CGM for patients with diabetes who require daily insulin therapy , unless they meet special criteria such as having hypoglycemia or inability to monitor glucose via traditional FSBGM.

Objectives Primary Study Aim: Among veterans with uncontrolled diabetes not requiring insulin therapy who are participating in an intensive multidisciplinary program to improve diabetes control (VDOP), to assess whether use of a CGM compared to use of traditional FSBGM results in greater change in hemoglobin A1c upon VDOP completion and up to 12 months.

Secondary study aims: To assess whether use of CGM in this population leads to greater improvement in diet, physical activity, and weight loss upon VDOP completion and up to 12 months.

Hypothesis

The use of a CGM by Veterans with T2DM who do not use insulin will help them improve their diabetes self - management (diet, physical activity, weight) and glycemic control more so than those using traditional fingerstick glucose monitoring.

Methods

This will be a prospective "open label" randomized controlled trial where participants will be randomly assigned to CGM (intervention group) or FSBGM (control group) during their participation in VDOP.

Relevance to Veterans and VA mission

Most Veterans with T2DM do not use insulin. It is important for both, these Veterans and the VA, to learn whether this more costly and somewhat burdensome technology supports improvement in diabetes self-management

ELIGIBILITY:
Inclusion Criteria:

* Successfully enrolled and ready to begin the VDOP program not on insulin therapy
* Type 2 diabetes by clinical history
* HbA1C between 8.0-12.0% inclusive within 3 months of enrollment
* Assessment by clinician that patient is willing to and able to wear a CGM device
* Stable diabetes medication regimen during the 3 months prior to entry

Exclusion Criteria:

* Patients already or planned on starting insulin therapy, already on CGM, or those who qualify for CGM under VA policy
* Patients with gestational diabetes or pregnant at time of screening or are planning to become pregnant during the study
* Patients with end stage renal disease (ESRD) on dialysis
* Anticipated acute uses of glucocorticoids (oral, injectable, or IV)
* Acute conditions that impact the HbA1c measurement stability such as GI blood loss, recent (within 3 months of study entry), anticipated red blood cell transfusion or erythropoietin administration
* Known or suspected significant allergy to use the Dexcom sensors
* Planning or currently enrolled on different weight program different from MOVE!
* Participating other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Glycemic Control | 12 months
  HbA1c

SECONDARY OUTCOMES:
Weight loss | 12 months
  lbs, Kg, and BMI

IPD SHARING:
Plan to Share IPD: No